CLINICAL TRIAL: NCT02221440
Title: Prophylactic Maternal Low Flow Nasal Oxygen Administration During the Second Stage of Labor for Fetal Distress
Brief Title: Maternal Oxygen Administration for Fetal Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Yunhai Chuai, Department of Obstetrics and Gynecology, Navy General Hospital, Beijing, Navy General Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CYH001
Record Dates: First submitted 2014-08-16; First posted 2014-08-20 (Estimated); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Oxygen Inhalation Therapy; Second Stage of Labour; Fetal Distress
MeSH Terms: conditions — Fetal Distress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- air, second stage of labor (Placebo Comparator): Patients randomized to the group will receive sham administered by nasal catheter.
  The therapy will continue until after delivery
  Interventions: Device: Low flow room air
- oxygen, second stage of labor (Experimental): Patients randomized to the group will receive oxygen administered by low flow nasal oxygen at a flow rate of 2 L/min.
  The therapy will continue until after delivery
  Interventions: Device: Low flow nasal oxygen

INTERVENTIONS:
Device: Low flow nasal oxygen — Oxygen will be administered by nasal catheter at a flow rate of 2 L/min. The therapy will continue until after delivery
  Arms: oxygen, second stage of labor
Device: Low flow room air — Sham: oxygen will be administered by nasal catheter at a flow rate of 0 L/min.
  Arms: air, second stage of labor

SUMMARY:
Supplementary oxygen is routinely administered to patients, even those with adequate oxygen saturations, in the belief that it increases oxygen delivery. However, oxygen delivery depends not just on arterial oxygen content but also on perfusion.

Maternal oxygen administration has been used in an attempt to lessen fetal distress by increasing the available oxygen from the mother. However, the effect of supplemental maternal oxygen therapy on fetal acid base status has been debated for more than seven decades.

Hypothesis: Prophylactic maternal low flow nasal oxygen administration during the second stage of labor can relieve fetal distress.

DETAILED DESCRIPTION:
A report from the cochran library (Cochrane Database Syst Rev. 2012 Dec 12;12:CD000136.):

Too little evidence to show whether oxygen administration to the woman during labour is beneficial to the baby.

Some babies show signs of distress, such as unusual heart rates or the passing of a bowel motion (meconium) during their mother's labour. This may be caused by a lack of oxygen passing from the woman to the baby through the placenta. Sometimes, women may be encouraged to breathe extra oxygen through a facemask (oxygen administration) to increase the oxygen available to the unborn baby. A review of two trials found too little evidence to show whether oxygen administration to the woman during the second stage of labour is beneficial to the baby. No trials of oxygen administration when the baby is showing signs of distress were found. Further research is needed.

ELIGIBILITY:
Inclusion Criteria:

* at term
* singleton
* primigraida
* cephalic presentation
* spontaneous or induced labor
* normal labor
* normal FHR tracings in the first stage
* at the onset of second stage

Exclusion Criteria:

* respiratory disease
* cardiovascular disease
* diabetes mellitus or insulin-treated gestational diabetes mellitus
* hypertension or preeclampsia
* oligohydramnios
* fetal growth restriction
* placental abruption
* anemia
* disorders in oxygen saturations
* received oxygen therapy in the first stage

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 443 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
cord arterial pH values (hydrogen ion concentration) less than 7.2 | within 30-60 seconds of birth
  Immediately after delivery (within 30-60 seconds of birth), umbilical cord arterial blood gas sample will be obtained.

SECONDARY OUTCOMES:
Apgar score less than 7 | at one and five minutes after birth
  The Apgar scale is determined by evaluating the newborn baby on five simple criteria on a scale from 0 to 2, then summing up the five values thus obtained. The resulting Apgar score ranges from 0 to 10. The five criteria are summarized using words chosen to form a backronym (Appearance, Pulse, Grimace, Activity, Respiration). The infant is given a score of 0, 1 or 2. The scores are added up and the total sum is their Apgar score.
  The test is generally done at one and five minutes after birth, and may be repeated later if the score is and remains low. Scores 7 and above are generally normal, 4 to 6 fairly low, and 3 and below are generally regarded as critically low.
maternal radial arterial partial pressure of oxygen | within 30-60 seconds of birth
  Immediately after delivery (within 30-60 seconds of birth), radial artery blood gas sample will be obtained.
umbilical cord venous partial pressure of oxygen | within 30-60 seconds of birth
  Immediately after delivery (within 30-60 seconds of birth), umbilical cord venous blood gas sample will be obtained.

OTHER OUTCOMES:
cesarean delivery rate | during the second stage of labor
assisted vaginal delivery | during the second stage of labor
maternal dissatisfaction | during the second stage of labor
abnormal fetal heart rate tracing | during the second stage of labor
neonatal resuscitation | within 10 mins of birth
neonatal encephalopathy | within 24 hours of birth
serious neonatal morbidity or death | within 28 days of birth

CONTACTS AND LOCATIONS:
Overall Officials: Yunhai Chuai, Dr, Principal Investigator — Navy General Hospital, Beijing
Locations (3):
- China (3):
  - Department of Obstetrics and Gynecology, Navy General Hospital., Beijing, Beijing Municipality
  - Navy General Hospital, Beijing, Beijing Municipality
  - Department of Obstetrics and Gynecology, Navy General Hospital., Beijing

REFERENCES:
- [Result] Qian G, Xu X, Chen L, Xia S, Wang A, Chuai Y, Jiang W. The effect of maternal low flow oxygen administration during the second stage of labour on umbilical cord artery pH: a randomised controlled trial. BJOG. 2017 Mar;124(4):678-685. doi: 10.1111/1471-0528.14418. PMID 28224745
- [Derived] Chuai Y, Jiang W, Xu X, Wang A, Yao Y, Chen L. Maternal oxygen exposure may not change umbilical cord venous partial pressure of oxygen: non-random, paired venous and arterial samples from a randomised controlled trial. BMC Pregnancy Childbirth. 2020 Sep 4;20(1):510. doi: 10.1186/s12884-020-03212-3. PMID 32887557